CLINICAL TRIAL: NCT00433342
Title: Study on the Effect of Flucloxacillin on the Serum Level of P-cresol in Peritoneal Dialysis Patients
Brief Title: The Effect of Antimicrobial Therapy on the Serum Level of P-cresol in Peritoneal Dialysis Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Björn Meijers, Dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML3532
Record Dates: First submitted 2007-02-07; First posted 2007-02-09 (Estimated); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Chronic Kidney Disease
Keywords: Antibiotic; p-cresol; peritoneal dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Floxacillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Flucloxacillin
  Interventions: Drug: Flucloxacillin
- II (No Intervention)

INTERVENTIONS:
Drug: Flucloxacillin — 500 mg QD oral
  Other Names: Floxapen
  Arms: I

SUMMARY:
An important subgroup of protein-bound toxins are generated as a result of protein fermentation in the colon. P-cresol is a fermentation metabolite of tyrosine. In renal failure, the colonic generation rate of p-cresol is markedly elevated. After absorption, the majority of p-cresol is conjugated to form p-cresyl sulphate. There is clear evidence, both in vitro and in vivo, that accumulation of conjugated fermentation metabolites is correlated with clinical important endpoints. Free p-cresol is an independent predictor for mortality in hemodialysis patients.

Moreover, in renal failure patients, neither hemodialysis nor peritoneal dialysis is capable of normalising the clearly elevated serum concentrations of p-cresyl sulphate. Removal is at least partially diminished by the important protein binding of p-cresol. Besides adaptation of renal replacement therapies to improve removal of protein bound solutes, another approach is to lower the generation of uremic toxins.

The mechanisms underlying colonic carbohydrate and protein fermentation, responsible for the generation of p-cresol, are only partially understood. On the one hand, the ratio of fermentable carbohydrates to proteins has been shown to be an important determinant of protein fermentation. On the other hand, changes in the colonic bacterial flora influence the generation of p-cresol in dogs and in healthy human individuals.

The effect of antibiotic therapy on bacterial protein fermentation and thus on the generation of p-cresol is not known. A reanalysis of data abstracted from a recent longitudinal study in peritoneal dialysis (PD) patients suggests that antibiotic therapy may lower p-cresol levels substantially. The current study aims at confirming these data in a prospective manner.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Exit site infection, requiring antibiotic treatment
* Maintenance therapy with peritoneal dialysis

Exclusion Criteria:

* Signs of peritonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-03; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
p-cresol reduction rate | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Björn Meijers, MD, Study Chair — UZ Leuven; Pieter Evenepoel, MD, PhD, Study Director — UZ Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Background] Bammens B, Evenepoel P, Keuleers H, Verbeke K, Vanrenterghem Y. Free serum concentrations of the protein-bound retention solute p-cresol predict mortality in hemodialysis patients. Kidney Int. 2006 Mar;69(6):1081-7. doi: 10.1038/sj.ki.5000115. PMID 16421516